CLINICAL TRIAL: NCT03065296
Title: Standardized Home Exercise Prescription: Education of Family Medicine Residents
Brief Title: Standardized Home Exercise Prescription Education
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Investigator left the institution and was withdrarwn
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB201602626
Record Dates: First submitted 2017-02-17; First posted 2017-02-27 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Behavior; Knowledge, Attitudes, Practice
Keywords: Behavior; education; medical residents; knowledge; confidence; skills assessment
MeSH Terms: conditions — Behavior | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Musculoskeletal (MSK) Exercise Prescription (Experimental): * Phase I: Residents will be surveyed as to their knowledge and confidence in both diagnosing specific musculoskeletal (MSK) issues and prescribing the correct home rehabilitation regimen.
  * In between phase 1 and phase 2 there will be a series of didactic lectures to educate resident on home exercise prescription and get them familiarized with the handouts.
  * Phase II: Residents will be surveyed again in May 2017 with the same multiple choice questions and Likert style confidence scales from phase 1
  The survey will consist of multiple choice and short essay questions, focused on the most common musculoskeletal (MSK) injuries seen in the primary care setting.
  Interventions: Behavioral: Musculoskeletal (MSK) Prescription Didactic Lectures; Other: Musculoskeletal (MSK) home exercise hand-outs

INTERVENTIONS:
Behavioral: Musculoskeletal (MSK) Prescription Didactic Lectures — In between phase 1 and phase 2 there will be a series of didactic lectures to educate resident on home exercise prescription and get them familiarized with the handouts.
Other: Musculoskeletal (MSK) home exercise hand-outs — In between phase 1 and phase 2, residents will use home exercise hand-outs readily available and educate their patients in regards to those.

SUMMARY:
This project will encompass an evaluation of the educational value of having evidence based home exercise protocols available for family medicine residents in regard to the prescription of home exercise treatment for common musculoskeletal conditions. Investigators will be evaluating resident knowledge on home exercise prescription as well as their level of comfort in educating their patients before and after a series of didactic sessions and implementation of exercise protocols.

DETAILED DESCRIPTION:
This study aims to fill the gap in this area of the literature pertaining to home exercise prescription. The justification of this study's scientific merit comes from the lack of literature and the need for research in this area. There have been multiple studies that have shown different exercise modality treatments for common musculoskeletal (MSK) complaints significantly improve both disability and overall quality of life. Despite the evidence of the short and long term effectiveness of exercise based therapies, there is a general lack of confidence of residents in prescribing and teaching patients rehab exercises.Additionally, many of the patients seen in the University of Florida (UF) Family medicine residency program cannot afford or do not have time to attend physical therapist led rehab sessions. This makes physician led education and the ability of prescribing exercise based treatments for musculoskeletal (MSK) complaints a very important component of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the Family Medicine Department at the University of Florida.

Exclusion Criteria:

* None

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in knowledge about Musculoskeletal (MSK) Exercises | at 6 months
  Knowledge scores should be at least overall 80% regarding MSK rehabilitation exercises.
Confidence in educating patients about Musculoskeletal (MSK) Exercises | at 6 months
  Improvement of at least 20% in Medical Residents' confidence regarding education of Musculoskeletal (MSK) to patients

SECONDARY OUTCOMES:
Confidence in prescribing Musculoskeletal (MSK) Exercises to patients | at 6 months
  Improvement of at least 20% in Medical Residents' confidence regarding prescription of Musculoskeletal (MSK) exercises
Improvement in prescribing Musculoskeletal (MSK) Exercises to patients | at 6 months
  Prescription scores should be at least overall 80% regarding MSK rehabilitation exercises

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Michaudet, MD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared.